CLINICAL TRIAL: NCT02639949
Title: The Use of Random Telephone Calls to Measure Immunosuppressive Therapy Adherence in Patients With Renal Transplants
Brief Title: Measuring and Improving Medication Adherence in Kidney Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: NIDDK_KUH
Record Dates: First submitted 2015-12-17; First posted 2015-12-28 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Kidney Transplant Recipients
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group CBT (Experimental)
  Interventions: Behavioral: Cognitive-behavioral adherence promotion program
- Standard Care (Active Comparator)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Cognitive-behavioral adherence promotion program — A culturally sensitive group cognitive behavioral therapy combined with adherence promotion.
  Arms: Group CBT
Behavioral: Standard Care
  Arms: Standard Care

SUMMARY:
Nonadherence to medication is a major obstacle to successful treatment of renal transplant patients. This study has two primary aims. The first is to test whether a culturally sensitive cognitive-behavioral adherence promotion program could significantly improve medication adherence to tacrolimus prescription. Participants will be randomly assigned to either group CBT or to standard care. The second aim is to pilot a novel strategy of adherence measurement - unannounced telephone pill counts, which has been shown to be a valid and reliable means to measure medication adherence in other patient populations. Participants will be recruited from waiting area of the kidney transplant clinic at SUNY Downstate Medical Center in Brooklyn, NY. Three unannounced telephone pill counts will be conducted prior to start of the intervention in order to establish baseline adherence and three pill counts will be conducted post-intervention. Tacrolimus trough concentration levels will also be collected as an additional biological measure of adherence.

ELIGIBILITY:
Inclusion Criteria:

- current prescription of tacrolimus less than 98% adherence to medication prescription as determined by three baseline pill counts

Exclusion Criteria:

- lack of telephone to complete pill counts lack of English proficiency to participate in adherence promotion sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Adherence as measured by unannounced telephone pill count | 3 months

SECONDARY OUTCOMES:
degree of agreement between pill count data and laboratory tacrolimus levels | 3 months

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829